CLINICAL TRIAL: NCT06203483
Title: The Comparison Of Ultrasound Guıded Adductor Canal Block And Perıcapsular Nerve Group Block For Postoperatıve Analgesıa Management Following Knee Arthroplasty Surgery
Brief Title: Ultrasound Guıded Adductor Canal Block vs Perıcapsular Nerve Group Block in Knee Artroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Mursel Ekinci, Assoc Prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa City Hospital 6
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Knee Disease; Knee Osteoarthritis; Knee Arthropathy
Keywords: Total Knee Arthroplasty; Postoperative Analgesia Management; Adductor Canal Block; Perıcapsular Nerve Group Block
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: There are two models for this study. Adductor canal block group, and pericapsular nerve group block group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor who performs postoperative pain evaluation will not know the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor canal block (Active Comparator): Adductor canal block will be performed at the end of the surgery. Patients will be administered tenoxicam (Tilcotil 20 mg flakon) 20 mg IV every 12 hours in the postoperative period. A patient controlled device prepared with 5 mg/ ml tramadol (100 mg-Contramal ® ampul) will be attached to all patients with a protocol included 10 mg bolus without infusion dose, 20 min lockout time and 4 hour limit. If the VAS score will be ≥ 4, 0,5 mg/kg-1 meperidine (Aldolan ampul 100 mg/2 ml) IV will be administered.
  Interventions: Drug: Adductor canal block
- PENG block (Active Comparator): PENG Block will be performed at the end of the surgery. Patients will be administered tenoxicam (Tilcotil 20 mg flakon) 20 mg IV every 12 hours in the postoperative period. A patient controlled device prepared with 5 mg/ ml tramadol (100 mg-Contramal ® ampul) will be attached to all patients with a protocol included 10 mg bolus without infusion dose, 20 min lockout time and 4 hour limit. If the VAS score will be ≥ 4, 0,5 mg/kg-1 meperidine (Aldolan ampul 100 mg/2 ml) IV will be administered.
  Interventions: Drug: PENG block

INTERVENTIONS:
Drug: Adductor canal block — A linear ultrasound probe will be placed medial to the patella, the probe will be advanced to cephalad, and the superficial femoral artery will be visualized. The block site will be confirmed by injecting 5 ml of saline around the saphenous nerve in the subsartorial region under ultrasound guidance. Then, 30 ml of local anesthetic solution containing 0.25% bupivacaine (Marcain 0.5% AstraZeneca, England) will be administered.
  Arms: Adductor canal block
Drug: PENG block — The probe will be placed at the anterior superior level of spina iliaca, parallel to the inguinal ligament. The probe will be scanned gradually towards the caudal. After the anterior inferior of the spina iliaca is visible, the probe will be slightly turned medially until the hyperechoic shadow of the superior pubic ramus is visible. The psoas muscle tendon will be visualized above the superior pubic ramus, then 5 ml of saline will be injected under the psoas tendon and the block location will be confirmed. After that 30 ml of 0.25% bupivacaine will be administered.
  Arms: PENG block

SUMMARY:
Knee arthroplasty surgery numbers are increasing depending on joint deformities and cartilage degenerations. Severe postoperative pain may occur in these patients due to surgery and the placed prosthesis.

The aim of study is to compare the effectiveness of AKB and PENG block for postoperative analgesia management after knee arthroplasty.

DETAILED DESCRIPTION:
Knee arthroplasty surgery numbers are increasing depending on joint deformities and cartilage degenerations. Severe postoperative pain may occur in these patients due to surgery and the placed prosthesis. Postoperative analgesia is important for early mobilization. So that, early movement of the joint is ensured and complications such as thromboembolism and infection are prevented. Various methods can be used for postoperative analgesia. One of these methods is epidural analgesia. However, it may not be applied due to the patient's refusal or the technical difficulties in the application. Another option is opioid agents. However; opioids have side effects such as nausea, vomiting, sedation, respiratory depression. Femoral nerve blockade can be done, but it is not preferred because it may prevent mobilization as a result of motor blockade.

Current regional anesthesia techniques used in knee surgery include selective blockade of the saphenous nerve in the adductor canal (adductor canal block-ACB) and pericapsular nerve group block (PENG). Adductor canal block; affects the vastus medialis branch of the saphenous nerve, one of the two largest sensory nerves from the femoral nerve to the knee, and the articular branches of the obturator nerve. Since the block is made in the distal thigh, the innervation of the quadriceps muscle is not affected, and therefore the motor power of this muscle is largely preserved. Another lower extremity peripheral regional blockade technique that is gaining importance today is PENG block. PENG, which is a musculofacial plane block made between the tendon of the psoas muscle and the ramus pubis, provides block of the femoral nerve, obturator nerve and accessory obturator nerve. In both block methods, pure sensory blockade provides analgesia without quadriceps muscle weakness, and this provides a significant advantage in terms of early mobilization.

The aim of this study is to compare these two analgesic methods in terms of effectiveness for postoperative analgesia management after knee arthroplasty. The primary outcome is to compare global recovery scores (QoR-15 scale), the secondary outcome is to compare postoperative pain scores (NRS), to evaluate postoperative opioid consumption, postoperative rescue analgesic (opioid) use, presence of motor blockade, postoperative first mobilization time, and side effects (allergic reaction, nausea, vomiting) associated with opioid use in this study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for total knee arthroplasty under spinal anesthesia

Exclusion Criteria:

* history of bleeding diathesis
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedur

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Global recovery scoring system (patient satisfaction scale) | The quality of recovery will be evaluated out of a total of 150 points according to the QoR-15 test to be applied at the portoperative 24th hour.
  The investigators will use the Turkish version of Quality of Recovery / QoR-15 questionairre
  PART A How have you been feeling in the last 24 hours? (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent])
  1. Able to breathe easily
  2. Been able to enjoy food
  3. Feeling rested
  4. Have had a good sleep
  5. Able to look after personal toilet and hygiene unaided
  6. Able to communicate with
  7. Getting support from hospital doctors and nurses
  8. Able to return to work or usual home activities
  9. Feeling comfortable and in control
  10. Having a feeling of general well-being
      PART B Have you had any of the following in the last 24 hours? (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor])
  11. Moderate pain
  12. Severe pain
  13. Nausea or vomiting
  14. Feeling worried or anxious
  15. Feeling sad or depressed

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | Patients will be evaluated at the first 24 hours period postoperatively.
  Postoperative 24 hours period. Patients' pain scores will be questioned at 0, 2, 4, 8, 16 and 24 hours.
The use of rescue analgesia | Meperidine consumption will be recorded at the first 24 hours period postoperatively.
  The need for rescue analgesia will be recorded at the first 24 hours period postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Mürsel Ekinci, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share IPD

REFERENCES:
- [Background] Kim S, Bosque J, Meehan JP, Jamali A, Marder R. Increase in outpatient knee arthroscopy in the United States: a comparison of National Surveys of Ambulatory Surgery, 1996 and 2006. J Bone Joint Surg Am. 2011 Jun 1;93(11):994-1000. doi: 10.2106/JBJS.I.01618. PMID 21531866
- [Background] Jiang X, Wang QQ, Wu CA, Tian W. Analgesic Efficacy of Adductor Canal Block in Total Knee Arthroplasty: A Meta-analysis and Systematic Review. Orthop Surg. 2016 Aug;8(3):294-300. doi: 10.1111/os.12268. PMID 27627711
- [Background] Kapoor R, Adhikary SD, Siefring C, McQuillan PM. The saphenous nerve and its relationship to the nerve to the vastus medialis in and around the adductor canal: an anatomical study. Acta Anaesthesiol Scand. 2012 Mar;56(3):365-7. doi: 10.1111/j.1399-6576.2011.02645.x. PMID 22335278
- [Background] Sahoo RK, Jadon A, Sharma SK, Nair AS. Pericapsular nerve group (PENG) block for hip fractures: Another weapon in the armamentarium of anesthesiologists. J Anaesthesiol Clin Pharmacol. 2021 Apr-Jun;37(2):295-296. doi: 10.4103/joacp.JOACP_295_20. Epub 2021 Jul 15. No abstract available. PMID 34349384
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251